CLINICAL TRIAL: NCT02235818
Title: Immediate Effectiveness of Counterforce Bracing Versus Kinesiotaping During Activity: A Randomized Crossover Trial in Patients With Lateral Epicondylosis
Brief Title: Determining the Immediate Effects of Counterforce Bracing Versus Kinesiotaping in Patients With Tennis Elbow
Acronym: LE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Joy MacDermid, Co-Director HULC Clinical Research lab, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSREB103099
Record Dates: First submitted 2013-07-04; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Tennis Elbow
Keywords: tennis elbow, treatment, lateral epicondylitis, immediate effects
MeSH Terms: conditions — Tennis Elbow | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesiotape (KT) (Active Comparator): Kinesiotape was used only on the affected side as per the manufacturer instructions. With the elbow extended, wrist fully flexed and fingers pointed down 24, KT was applied with slight stretch (10-15%) and paper off tension to the lateral arm beginning just above the bony portion of lateral epicondyle. Once the top strand was anchored, KT was applied along the side of elbow such that hole in the tape was over lateral epicondyle of the elbow. Two strands of tape followed the lateral forearm and ended at around beginning of the distal one third of forearm. Once the support was applied, KT was gently rubbed to activate the glue.
  Interventions: Device: Kinesiotape
- Counterforce elbow brace (Active Comparator): The counterforce brace was approximately 5cm wide with velcro attachment for adjustable girth. It had gel pack for extra support on extensor muscle mass. With the elbow extended, brace was applied 2.5cms below the lateral epicondyle. A feeling of comfortable compression, as reported by the patients was used to adjust the brace.
  Interventions: Device: Counterforce elbow brace

INTERVENTIONS:
Device: Kinesiotape — Pre-cut kinesiotape for tennis elbow, spidertech.com, applied on wrist extensors starting above elbow and ending at distal one third of forearm
  Other Names: elastic tape, elastic therapeutic tape, kinesiotex tape
  Arms: Kinesiotape (KT)
Device: Counterforce elbow brace — Applied over the wrist extensor muscle mass, had velcro for adjustment, comfortable grip as reported by patient was used to adjust the brace
  Other Names: elbow strap, forearm brace, forearm strap
  Arms: Counterforce elbow brace

SUMMARY:
The purpose of this study was to compare the immediate efficacy of Counterforce brace versus kinesiotaping on patients with lateral epicondylosis/tennis elbow with respect to a repetitive physical task. The investigators hypothesized that there would be difference in the outcomes with respect to interventions and activity. Patient came for one hour long Single occasion testing session and were not followed up after the testing was complete.

DETAILED DESCRIPTION:
This was a cross over randomized control trial. Thirty patients with clinical diagnosis of lateral epicondylosis/tennis elbow were recruited from a local community and were tested on single occasion (one time testing session) before and after a five minute upper extremity repetitive task first with control and then brace and kinesiotape assigned in cross-over design. The testing session was one hour long and there was no follow up of patients following the testing. The patients were recruited between Jan-June 2013.

ELIGIBILITY:
Inclusion Criteria:

1. Age (18-70 years)
2. Ability to provide written informed consent to participate
3. Were at least three weeks from onset of symptoms
4. Complaints of discomfort or pain at the lateral elbow region for a minimum of three weeks and tenderness with palpation of the lateral epicondyle
5. Provocation of lateral elbow pain with one of the following test - resisted middle finger extension, resisted wrist extension or passive stretch of wrist extensors

Exclusion Criteria:

1. History of surgery on affected elbow
2. History of cortisone injections on the affected elbow in the past 4 weeks
3. Any physical or mental limitations that precluded performance of the study testing
4. Allergy to adhesive tapes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pain free grip strength | initial visit
  Pain free grip strength was recorded with J-tech medical dynamometer before and after five minutes of repetitive physical exposure with first control (no intervention) and then brace and kinesiotape assigned randomly in cross-over fashion.

SECONDARY OUTCOMES:
Pressure Pain Threshold | initial visit
  Pressure Pain Threshold was recorded with J-tech medical Algometer before and after five minutes of repetitive physical exposure with first control (no intervention) and then brace and kinesiotape assigned randomly in cross-over fashion.

OTHER OUTCOMES:
Pain levels | initial visit
  Pain levels were recorded with Numeric Pain Rating scale before and after five minutes of repetitive physical exposure with first control (no intervention) and then brace and kinesiotape assigned randomly in cross-over fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Joy C Macdermid, PT, PhD, Principal Investigator — Western University, Canada; Pritika Gogia, MSc, Principal Investigator — Western University, Canada
Locations (1):
- The Hand and Upper Limb Centre, St. Joseph's Health Centre, London, Ontario, Canada